CLINICAL TRIAL: NCT05510401
Title: Multicenter Clinical Investigation for the Evaluation of Safe Use of SECURIDRAP® SELFIA®
Brief Title: Evaluation of Safe Use of SECURIDRAP® SELFIA®
Acronym: SECURIDRAP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Groupe Mulliez-Flory (Industry)
Collaborators: EVAMED (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2019-A03234-53
Record Dates: First submitted 2022-03-07; First posted 2022-08-22 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Disorientation; Cognitive Impairment; Behavior Disorders
Keywords: disorientation; nocturnal behavioral disorders; major cognitive impairment
MeSH Terms: conditions — Confusion; Cognitive Dysfunction; Mental Disorders

STUDY DESIGN:
Intervention Model Description: non-comparative clinical investigation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SECURIDRAP® SELFIA® (Other): Use of a SECURIDRAP® SELFIA® restraint system Monitoring with passage of an independent assessor
  Interventions: Other: SECURIDRAP® SELFIA®

INTERVENTIONS:
Other: SECURIDRAP® SELFIA® — Use of SECURIDRAP® SELFIA® for 15 night

SUMMARY:
Interventional, multicenter, prospective and non-comparative clinical investigation carried out in 9 French establishments in order to assess the safety of the SÉCURIDRAP® SELFIA® bedding by mesasuring all the adverse events likend to its use.

Following the withdrawal from the market of the first version of the SECURIDRAP® SELFIA®, this clinical investigation is being carried out at the request and on the recommandation of the ASNM in order to assess the safety of the second version of the SECURIDRAP® SELFIA® coating.

DETAILED DESCRIPTION:
The proposed study is a prospective, multicenter, interventional and non-comparative research.

This clinical investigation is carried out in real life in accordance with the usual care for all patient with a prescription for SECURIDRAP® SELFIA® and who meet the eligibility criteria, in nursing homes and public and private hospitals based in France.

This interventional clinical investigation with minimal risks and constraints aims to confirm the safety of use of SECURIDRAP® SELFIA® in healthcare establishment.

The patient will be followed for 15 nigths, during witch an independent assessor will ensure that the conditions of use os the SECURIDRAP® SELFIA® sleeping bag are respected.

ELIGIBILITY:
Inclusion Criteria:

* Patient at least 18 years old
* Patient having a medical prescription for SÉCURIDRAP® SELFIA®
* Patient in phase or state of disorientation
* Patient with nocturnal behavior disordre
* Patient with major cognitive impairment
* Patient at risk of falling into bed
* Patient subject to guardianship or curatorship
* Patient beneficiary or affiliated to a social security scheme
* Patient who has given their participation agreement aand informed consent

Exclusion Criteria:

* Patient and/or guardianship or curatorship refusing to agree to participate in the clinical investigation
* Patient in psychiatry
* Patient with severe agitation
* Patient who will be agitated once installed in the SÉCURIDRAP® SELFIA®
* Patient with intolerance to the medical device
* Patient able to extract himself from SÉCURIDRAP® SELFIA®
* Patient able to unlock the bed rails by himself
* Patient without social coverage or not benefiting from it through a third party
* Patient minor, pregnant woman, persons deprived of their liberty
* Patient who participating or having participated in another clinical investigation, drug or medical device in the 30 days preceding inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2022-05-18 (Actual); Primary Completion 2025-03-30 (Estimated); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
Rate of occurrence of adverse events related to the use of SÉCURIDRAP® SELFIA® | [15 days]
  quotient of the number of overnight stays or at least one adverse event related to the use of SÉCURIDRAP® SELFIA® appeared, by the number of overnight stays where SÉCURIDRAP® SELFIA® was used

SECONDARY OUTCOMES:
Rate of occurrence of user errors that could endanger patient safety | [15 days]
  These usage errors will be measured during the verification of correct use of the SÉCURIDRAP® SELFIA® by the independent assessor, 2 hours after patient has been installed in the medical device
Rate of patients remaining bedridden each night for the duration of the sudy | [15 days]
  P = [(NNL)/ (NU)] x 100 with:
  * NNL : the number of nights , patient has not released
  * NU : the number of use; (number of overnight stays)
Satisfaction rate of healthcare teams using SÉCURIDRAP® SELFIA®, in terms of time savings, weel-being, comfort and respect for the dignity of patient | [15 days]
  Time saving for healthcare teams via a graduated scale of 0-10 The weel-being / comfort of the patient via a graduated scale of 0-10 Respect for the dignity of the patient via a graduated scale of 0-10
The learning curve for using SECURIDRAP® SELFIA® by healthcare team | [15 days]
  The curve reflects the time required for nursing expertise in the use of SECURIDRAP.

CONTACTS AND LOCATIONS:
Overall Officials: François Pr PUISIEUX, Principal Investigator — CHU Lille; Aline Dr CORVOL, Principal Investigator — CHU Rennes; Sabine Dr AHMINE, Principal Investigator — Hospices Civils de Lyon; Thierry Dr LECRIQUE, Principal Investigator — CSSR La Clauze; Brigitte Dr GERS, Principal Investigator — USSAP- ASM LIMOUX; Marguerite Dr REY, Principal Investigator — USSAP- ASM LIMOUX; Valérie Dr WIEL, Principal Investigator — EHPAD l'Aquarelle; Brigitte Dr TILMONT, Principal Investigator — CMMF de Bailleul; Eddy Dr BAHEU, Principal Investigator — CH Hazebrouck; Denis Dr LEFEBVRE, Principal Investigator — CH Le Quesnoy; Philippe Dr VEAU, Principal Investigator — CSSR La Clauze; Pearlide Dr Kizonzolo-de-Bello, Principal Investigator — CHG Roubaix
Locations (10):
- France (10):
  - CMMF de Bailleul, Bailleul
  - EHPAD l'Aquarelle, Bully-les-Mines
  - Centre Hospitalier d'Hazebrouck, Hazebrouck
  - Centre Hospitalier Le Quesnoy, Le Quesnoy
  - CHU Lille, Lille
  - Ussap- Asm Limoux, Limoux
  - CHU Lyon, Lyon
  - CHU Rennes, Rennes
  - CHG Roubaix, Roubaix
  - CSSR La Clauze, Saint-Jean-Delnous

IPD SHARING:
Plan to Share IPD: No